CLINICAL TRIAL: NCT04206046
Title: The Effect of Regional Anaesthesia and Genetic Factors in the Development of Chronic Pain Following Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sciberras, Stephen M.D. (Individual)
Responsible Party: Principal Investigator, Stephen Sciberras, Lead investigator, Sciberras, Stephen M.D.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 001
Record Dates: First submitted 2019-12-12; First posted 2019-12-20 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Arthroplasty, Replacement, Knee; Chronic Pain Post-Proceduraal
Keywords: arthroplasty, knee; chronic pain
MeSH Terms: conditions — Chronic Pain | interventions — Anesthesia, Spinal; Anesthesia, General

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General Anaesthesia (Active Comparator): Patients will receive a general anaesthetic, together with a femoral nerve block.
  Interventions: Procedure: General anaesthesia
- Spinal Anaesthesia (Active Comparator): Patients will receive a spinal anaesthetic
  Interventions: Procedure: Spinal anaesthesia

INTERVENTIONS:
Procedure: Spinal anaesthesia — Patients will receive a spinal anaesthetic
  Arms: Spinal Anaesthesia
Procedure: General anaesthesia — patients will receive a general anaesthetic and a femoral nerve block
  Arms: General Anaesthesia

SUMMARY:
The study aims to assess the effect of spinal anaesthesia against a general anaesthesia with a femoral block, with respect to the incidence of chronic pain following a total knee replacement.

It will also focus on genetic factors and their influence on chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* patients able to undergo a total knee arthroplasty

Exclusion Criteria:

* age more than 75 years
* known case of chronic pain syndromes
* arthroplasty not due to osteoarthritis
* sensitivity to any drugs used in protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain Numerical Rating Scale on physiotherapy | 24 hours
  Pain Numerical Rating Scale, from 0 (no pain) to 10 (severe pain)
WOMAC Score at 3 and at 6 months | 6 months
  WOMAC score, ranging from 0 to 94
WOMAC Pain Score at 3 and at 6 months | 6 months
  WOMAC Pain score, ranging from 0 (no pain) to 20 (severe pain on numerous activities)

SECONDARY OUTCOMES:
Morphine consumption | 24 hours
  Morphine use postop
Pain Numerical Rating Scale after 6 months | 6 months
  Pain Numerical Rating Scale at rest, from 0 (no pain) to 10 (severe pain)
Incidence of Chronic Post-surgical Pain | 6 months
  WOMAC pain score greater than 5 at 6 months (out of total of 20)
Change in WOMAC Score at 3 and at 6 months | 6 months
  change in WOMAC score, ranging from 0 to 94
Change in WOMAC Pain Score at 3 and at 6 months | 6 months
  change in WOMAC Pain score, ranging from 0 (no pain) to 20 (severe pain on numerous activities)

CONTACTS AND LOCATIONS:
Locations (1):
- Mater Dei Hospital, Msida, Malta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sciberras SC, Vella AP, Vella B, Spiteri J, Mizzi C, Borg-Xuereb K, LaFerla G, Grech G, Sammut F. A randomized, controlled trial on the effect of anesthesia on chronic pain after total knee arthroplasty. Pain Manag. 2022 Sep;12(6):711-723. doi: 10.2217/pmt-2021-0081. Epub 2022 Mar 30. PMID 35350864

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/46/NCT04206046/Prot_SAP_000.pdf